CLINICAL TRIAL: NCT02908984
Title: Effects of Specific Neck Rehabilitation on Patients With Unilateral Headache and Neck Pain (Cervicogenic Headache), and Relation to Structural and Functional Changes in the Brain
Brief Title: Specific Neck Rehabilitation for Unilateral Headache and Neck Pain, and Structural and Functional Changes in the Brain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1652
Record Dates: First submitted 2016-01-14; First posted 2016-09-21 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Cervicogenic Headache
Keywords: unilateral headache; cervical pain; neck pain; rehabilitation; structural brain changes; surface based volumetry; diffusion tensor imaging; functional brain changes; sensorimotor control; craniocervical flexion; vestibular rehabilitation; cortical thickness
MeSH Terms: conditions — Post-Traumatic Headache; Headache; Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Specific neck rehabilitation (Experimental): The intervention includes specific neck rehabilitation as described by Jull and Falla over a period of 4 weeks and recommendations for further training.
  Interventions: Behavioral: Specific neck rehabilitation
- Standard primary health care (Active Comparator): This represents individualized therapy administered by the primary physician.
  Interventions: Other: Standard primary health care

INTERVENTIONS:
Behavioral: Specific neck rehabilitation — Guided craniocervical, axioscapular and proprioceptive training that includes education, postural exercises, as well as training of cervical and shoulder muscles, and vestibular rehabilitation, included oculomotor function if indicated, and general exercises
  Arms: Specific neck rehabilitation
Other: Standard primary health care — The treatment may include pharmacological medication, chiropractic and physiotherapy or no active treatment
  Arms: Standard primary health care

SUMMARY:
In part 1 of the project clinical effect of specific neck rehabilitation for unilateral headache and neck pain (also termed cervicogenic headache) will be compared with standard primary health care. The researchers will further study whether fear avoidance beliefs and self-efficacy predict long term neck function and headache frequency superior to active range of neck movement. Part 2 will investigate whether patients with cervicogenic headache have structural changes in cerebral grey and white matter and in connectivity of the resting state state network, and whether these are reversed after effective neck rehabilitation and correlate to symptom severity and degree of disability.

DETAILED DESCRIPTION:
The project includes two parts:

Part 1: With a longitudinal semicross-over, randomized control design the investigators will compare the clinical efficacy of a 6 month specific neck rehabilitation with standard primary health care on patients with unilateral headache and neck pain ( also termed cervicogenic headache) and study whether self-efficacy and fear avoidance beliefs predict 12 month self-reported neck function and headache frequency superior to the active range of neck movement The patients will either receive a specific neck rehabilitation program or 6 month standard primary health care before they cross over to neck rehabilitation. Sociodemographic and clinical characteristics will be collected before each treatment session and 6 and 12 months later.

Part 2: With a non-randomized comparative design including a subsample of the patients (n: 36) and healthy controls (n: 36) the investigators will explore whether there are structural changes in the cerebral grey and white matter, and whether cerebral connectivity within the default mode network (DMN and other major cerebral networks) are significantly different and whether the changes correlate to symptom severity and degree of disability.

Structural (cortical volume and thickness) changes will measured by volumetric magnetic resonance imaging (MRi) and diffusion tensor imaging (DTI), while cerebral connectivity by resting state fMRI (rs-fMRI). Whether the anticipated cerebral changes in volume, structure and connectivity are reversed after specific neck rehabilitation will be tested by repeated measurements. Analyses of MRI scans and clinical characteristics will be performed before each treatment session and 6 months later.

Statistics: A parallel design power calculations based on previous studies indicated that for the clinical part a number of 21 patients within each treatment group (a total of 42 patients) and for the MR analyses a subsample of 34 patients and 34 health controls will be sufficient to obtain a statistical power of 80% with a p-value of 5%. Given a 2:1 ratio following a semi-cross over design, normal distributed data, α = 0.05, different standard deviations for each group (SD 1,38 and 1,71), and a statistical power of 0,8, a calculation indicated a sample size of 36 patients for the RCT. With a dropout rate up to 35%, 54 participants would be satisfactory.

Changes between baseline and the 6 month follow up will be used for "between and within group" comparisons while 12 months data will be included for in "within-group" comparisons. Statistical predictor analyses will be performed by regression analyses. The statistician who are performing the primary end point analysis, are blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral headache and neck pain for 2 years or more
* Minimum one headache attack pr week (numeric rating scale ≥4)
* Five or more of Antonaci's seven diagnostic criteria
* Neck Disability Index score ≥8 Points (≥16 percent points).

For healthy controls:

• Same age distribution

Exclusion Criteria:

* Progressive diseases (rheumatoid arthritis, cancer)
* Ongoing cervical infection
* Neurological disease (syringomyelia, radiculopathy, multiple sclerosis, Parkinson's disease, ischemic stroke )
* Other headache (>1 tension type headache or migraine attack every month)
* Other pain conditions (including primary temporomandibular disorder and generalized pain (fibromyalgia with pain intensity >6 to digital palpation)
* Previous or ongoing drug abuse
* Serious psychiatric disorder.
* Hopkins Symptom Checklist-25 score for depressive symptoms > 2.2
* Ongoing litigation process
* Intolerance to MRI
* Pregnancy and lactation
* For the subsample undergoing MR analyses: Other systemic diseases (Hypertension, hyperlipidemia, diabetes mellitus, heart disease, cerebrovascular, epilepsy or other vascular diseases) and dysmenorrhea requiring analgesics

For healthy controls:

* Exclusion criteria as above
* Chronic pain
* Chronic dizziness
* Intolerance to MRI
* Pregnancy and lactation

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference of days with headache pr week after specific neck rehabilitation vs standard primary health care | 6 months after baseline
  Between group comparison with a numeric variable (scale 0-7)
Differences in grey matter volume of the brain and brain stem between patients with unilateral headache and neck pain vs. healthy controls | Baseline
  Two independent group comparison based on volumetric analysis of cerebral grey matter also including surface based measurements (continuous variable)
Differences in cortical thickness between patients with unilateral headache and neck pain vs. healthy controls | Baseline
  Two independent group comparison based on surface based analyses of cerebral grey matter carried out with FreeSurfer version 6.0

SECONDARY OUTCOMES:
Difference in pain intensity after specific neck rehabilitation vs. standard primary health care | 6 months after baseline
  Between group comparison with a numeric variable (scale 0-10)
Improved neck function after specific neck rehabilitation vs. standard primary health care | 6 months after baseline
  Between group comparison with a numeric variable (scale 0-50)
Change in grey matter volume of the brain and brain stem in patients with unilateral headache and neck pain after specific neck rehabilitation | 6 months
  Within group comparison based on volumetric analysis of cerebral grey matter also including surface based measurements (continuous variable)
Change in cortical thickness of the brain between patients with unilateral headache and neck pain after specific neck rehabilitation | 6 months
  Within group comparison based on surface based volumetric analysis of cerebral grey matter (continous variable)
Differences in white matter integrity in patients with unilateral headache and neck pain vs. healthy controls | Baseline
  Two independent group comparison based on diffusion tensor imaging with tract based spatial statistics analyses
Difference in white matter integrity after specific neck rehabilitation vs standard primary health care | 6 months after baseline
  Between group comparison based on diffusion tensor imaging with tract based spatial statistics analyses
How four week baseline headache intensity reported by a numeric rating scale is associated with regional grey matter volumes measured by surface based volumetry in patients with unilateral headache and neck pain. | Baseline
  Linear regression analysis will be performed where the surface based volumetric measure of cerebral grey matter is the dependent variable, and four week baseline headache intensity is independent variable. Baseline headache intensity is based on daily measures during the last 4 weeks and is reported by an electronic diary and numeric rating scale where 0 is no pain and 10 is worst imaginable pain. It is thus considered a continuous measure. Age and gender are included as covariates.
How baseline perceived cognitive function predicts volumetric differences of cerebral grey matter in patients with unilateral headache and neck pain | Baseline
  Linear regression analysis of surface based volumetric measures of grey matter (continuous data) and scores of Everyday Memory Questionnaire (scale 0-8).
How baseline active range of neck movement predicts neck function | 12 months after baseline
  A logistic regression analysis on how baseline active range of neck movement (continuous data, degrees of rotation) predicts a 30% reduction in Neck Disability Index Score (0-50). Co-factors are age, gender, education, sick-leave.
How baseline active range of neck movement predicts headache frequency | 12 months after baseline
  A logistic regression analysis on how baseline active range of neck movement (continuous data, degrees of rotation) predicts a 30% reduction in headache frequency (0-7). Co-factors are age, gender, education, sick-leave.
How baseline self efficacy predicts neck function | 12 months after baseline
  A logistic regression analysis on how baseline General self efficacy scale score (scale 10-40) predicts a 30% reduction in Neck Disability Index Score (0-50). Co-factors are age, gender, education, sick-leave.
How baseline self efficacy predicts headache frequency | 12 months after baseline
  A logistic regression analysis on how baseline General self efficacy scale score (scale 10-40) predicts a 30% reduction in headache frequency (0-7). Co-factors are age, gender, education, sick-leave.
How baseline fear avoidance beliefs for physical activity predict neck function | 12 months after baseline
  A logistic regression analysis on how baseline fear avoidance beliefs score predict a 30% reduction in Neck Disability Index Score (0-50). Co-factors are age, gender, education, sick-leave.
How baseline fear avoidance beliefs for physical activity predict headache frequency | 12 months after baseline
  A logistic regression analysis on how baseline fear avoidance beliefs for physical activity score predict a 30% reduction in headache frequency (0-7). Co-factors are age, gender, education, sick-leave.
Difference in intra-network connectivity of resting state networks in patients with unilateral headache and neck pain vs. healthy controls. | Baseline
  Two independent comparison based on baseline rs-fMRI data to compare patients and controls. In multivariate general linear models, the investigators will use DMN and other major cerebral networks, identified by independent component analysis (ICA), as dependent variables and test whether there are differences in cerebral connectivity between patients and controls. All rs-fMRI analyses will be performed with the GIFT software http://mialab.mrn.org/software/gift/index.html. An ICA procedure in GIFT will be used to identify functional networks. GIFT that has a MatLab based statistical module for general linear modelling (GLM) of rs-fMRI data that will be used for all rs-fMRI analyses.
Change of resting state connectivity in patients who report reduction in headache attacks. | 6 months after baseline
  Within group comparison of resting state networks between baseline and 6 months follow up in a repeated measure GLM in the GIFT. Connectivity of DMN and other major networks is dependent variable and change in number of headache attacks main predictor variable.
Changes of resting state connectivity related to pain relief after specific neck rehabilitation. | 6 months
  Within group comparison of resting state networks between baseline and 6 months follow up in a multivariate GLM. Change of connectiviy in DMN and other major networks is dependent variables and pain reports main covariate.
Changes in connectivity of resting state networks related to improved craniocervical flexion endurance capacity after specific neck rehabilitation. | 6 months
  Within group comparison of resting state networks between baseline and 6 months follow in a multivariate GLM. Connectivity of DMN and other major networks is dependent variables and craniocervical flexion endurance capacity main covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnvald Kvarstein, PhD, Principal Investigator — UiT The Arctic University of Tromsø
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No